CLINICAL TRIAL: NCT00229203
Title: "Phase II Multicenter, Open-Label, Clinical and Pharmacokinetic Study of Aplidin® As A 3-Hour Infusion Every 2 Weeks Alone or in Combination With Dexamethasone, in Pre-Treated Patients With Relapsing or Refractory Multiple Myeloma."
Brief Title: A Study of Aplidin (Plitidepsin) 3 h iv in Subjects With Relapsing or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: PharmaMar USA Inc., PharmaMar USA Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-014-03
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Aplidin; Plitidepsin; PharmaMar
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Plitidepsin — 3-hour infusion every 2 weeks alone or in combination with dexamethasone

SUMMARY:
This is a phase II study to determine the efficacy following treatment with Aplidin® 5 mg/m2, given as a 3 hours intravenous infusion every 2 weeks, in patients with relapsed or refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
This is a phase II study to determine the efficacy following treatment with Aplidin® 5 mg/m2, given as a 3 h iv infusion every 2 weeks, in patients with relapsed or refractory multiple myeloma (MM) and to obtain the following :

* Additional pharmacokinetic information for Aplidin® given as 3-hour IV infusion every 2 weeks in patients with MM.
* To obtain additional genomic and pharmacodynamics information on MM and Aplidin.
* To assess the safety and tolerability of Aplidin® given as 3-hour IV infusion every 2 weeks in patients with MM alone or in combination with dexamethasone given orally as a 20 mg daily for 4 days
* To determine the response rate in the second cohort of patients following treatment with Aplidin®, given as a 3 hour infusion every 2 weeks, plus dexamethasone given orally as a 20 mg daily for 4 days, starting the same day of Aplidin® administration, as a second treatment stage in patients with suboptimal response to Aplidin® as single agent (progressive disease after three cycles or stable disease after four cycles).

ELIGIBILITY:
Inclusion criteria

1. Written informed consent obtained from the patient before starting any study-specific procedure. If any patient is unable to give consent, it may be obtained from the patient's legal representative if in accordance with local laws and regulations
2. Age ≥ 18 years
3. Performance status Eastern Cooperative Oncology Group (ECOG) ≤ 2
4. Life expectancy ≥ 3 months.
5. Patient was previously diagnosed with MM based on standard criteria and currently requires treatment because MM relapses following a response to standard chemotherapy or high-dose chemotherapy, or MM is refractory (i.e., failure to achieve at least complete response (CR), partial response (PR) or stable disease (SD)) to their most recent chemotherapy.
6. Patient has measurable disease, defined as follows:

   * For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value and, where applicable, urine light-chain excretion of ≥ 200 mg/24 hours.
   * For oligo or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. Magnetic resonance imaging (MRI), Computerized Axial Tomography (CT-Scan)).
7. Recovery from any non-hematological toxicity derived from previous treatments. The presence of alopecia and National Cancer Institute Common Toxicity Criteria (NCI-CTC) grade < 2 sensitive peripheral neuropathy is allowed.
8. Patient has the following laboratory values within 14 days before day 1, cycle 1:

   * Platelet count ≥ 50 x109/L, hemoglobin ≥ 8.0 g/dl and absolute neutrophil count (ANC) ≥ 1.0x109/L; lower values may be accepted if clearly are due to bone marrow involvement by multiple myeloma.
   * Corrected serum calcium < 14mg/dL.
   * Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal.
   * Alanine transaminase (ALT): ≤ 2.5 x the upper limit of normal.
   * Total bilirubin: ≤ 1.5 x the upper limit of normal.
   * Calculated Creatinine clearance: ≥ 40 mL/minute (by means of Crockoft and Gault´s formula).
9. Left ventricular ejection fraction within normal limits.

Exclusion criteria

1. Prior therapy with Aplidin®.
2. Pregnant or lactating women; men and women of reproductive potential who are not using effective contraceptive methods (double barrier method, intrauterine device, oral contraception)
3. History of another neoplastic disease. The exceptions are:

   * non-melanoma skin cancer,
   * carcinoma in situ of uterine cervix,
   * any other cancer curatively treated and no evidence of disease for at least 10 years.
4. Other relevant diseases or adverse clinical conditions:

   * History or presence of unstable angina, myocardial infarction, valvular heart disease or congestive heart failure.
   * Previous mediastinal radiotherapy.
   * Uncontrolled arterial hypertension despite optimal medical therapy.
   * Previous treatment with doxorubicin at cumulative doses in excess of 400 mg/m².
   * Symptomatic arrhythmia or any arrhythmia requiring treatment.
   * History of significant neurological or psychiatric disorders
   * Active infection
   * Patient is known to be human immunodeficiency virus (HIV) positive, Hepatitis B surface antigen-positive or active hepatitis C infection.
   * Myopathy or any clinical situation that causes significant and persistent elevation of creatine kinase (CK)(>2.5 ULN in two different determinations performed with one week apart)
   * Significant non-neoplastic liver disease (e.g. cirrhosis, active chronic hepatitis)
   * Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months)
5. Limitation of the patient's ability to comply with the treatment or follow-up protocol.
6. Treatment with any investigational product in the 30 days period before inclusion in the study or radiotherapy in the 4 weeks before inclusion in the study. Other previous treatments should have been completed 3 weeks before inclusion in the study, and in case of high dose chemotherapy, 8 weeks.
7. Known hypersensitivity to Aplidin®, mannitol, cremophor, or ethanol or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Study Chair — Chief division hematological malignancies - Medical Oncology - Dana Farber Cancer Institute - Harvard Medical School, Boston
Locations (1):
- Jerome Lipper Multiple Myeloma Center - Dept of Medical Oncology - Dana Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in 10 centers in Spain and USA between June 2004 and June 2008.
Groups:
- Plitidepsin: Plitidepsin 5 mg/m2 given as a 3-hour i.v. infusion every two weeks.
- Plitidepsin + Dexamethasone: Plitidepsin 5 mg/m2 given as a 3-hour i.v. infusion every two weeks plus 20 mg of oral dexamethasone every day on days 1 to 4 of each cycle, starting at the same time than the plitidepsin infusion.
Period: Overall Study
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Started | 32 | 19
Completed | 0 | 0
Not Completed | 32 | 19
Not completed — Progressive disease | 18 | 9
Not completed — Toxicity | 6 | 1
Not completed — Death | 4 | 2
Not completed — Other | 3 | 3
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone | Total
Number analyzed (Participants) | 32 | 19 | 51
Age Continuous [Median (Full Range); unit: years] | 66 [47 to 82] | 63 [47 to 86] | 64.0 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 17 | 13 | 30
ECOG PS [Number; unit: patients] — ECOG PS: Eastern Cooperative Oncology Group Performance Status This scale is used by doctors to assess how a patient's disease is progressing, how the disease affects the daily living abilities of patients, and determine appropriate treatment and prognosis. Scale points: 0, 1, 2, 3, 4 & 5; 0: Fully active, able to carry on all pre-disease performance without restriction, and 5: Death
  patients
    0 Units of Scale | 6 | 6 | 12
    1 Units of Scale | 18 | 9 | 27
    2 Units of Scale | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Defined as the Combined Rate of Complete Response, Partial Response and Minimal Response
Description: Complete response(CR):0 percentage the original monoclonal protein level from blood and urine Partial response(PR): ≥50 percentage reduction in the level of serum monoclonal protein Minimal response(MR):≥25 percentage to ≤ 49 percentage reduction in the level of serum monoclonal protein Stable disease: Not meeting the criteria for MR or PD. Progressive disease: >25 percentage increase in level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation.
  Treatmen failure: Reappearance of serum or urinary paraprotein
Time Frame: Every 2 weeks until progression or death occurs.
Population: Per protocol - Only 29 of 32 and 18 of 19 enrolled patients were evaluable (analyzed patients)
Measure: Number; unit: percentage patients
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Number analyzed (Participants) | 29 | 18
percentage patients
  Complete response | 0 | 0
  Partial response | 3 | 11
  Minimal response | 7 | 11
  Stable Disease/No changes | 41 | 61
  Progressive Disease/Treatment failure | 48 | 17

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression (TTP):date of first infusion to the date of documented progressive disease which can be defined as >25 percentage increase in level of serum monoclonal paraprotein.
Time Frame: Every 2 weeks until progression or death due to progression occurs. Median TTP and TTP rates at 3 months and 6 months were assessed.
Population: Per protocol - Only 29 of 32 and 18 of 19 enrolled patients were evaluable (analyzed patients)
Measure: Median (Full Range); unit: months
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Number analyzed (Participants) | 29 | 18
months | 2.3 [1.5 to 2.8] | 4.2 [3.4 to 7.7]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS): time from the date of first infusion to the date of documented progression or death
Time Frame: Every 2 weeks until progression or death occurs. Median PFS and PFS rates at 3 months and 6 months were assessed.
Population: Per protocol - Only 21 of 32 and 8 of 19 enrolled patients were evaluable (analyzed patients)
Measure: Median (Full Range); unit: months
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Number analyzed (Participants) | 21 | 8
months | 2.3 [1.4 to 2.6] | 3.8 [3.1 to 7.7]

4. Secondary Outcome: Number of Patients With Overall Survival (OS)
Description: Overall Survival (OS): time from the date of first infusion to the date of documented death
Time Frame: Start of treatment to death. At each patient visit while on treatment, then every 3m during follow-up. Median OS and OS rates at 6 months and 12 months were assessed.
Population: Per protocol - Only 21 of 32 and 8 of 19 enrolled patients were evaluable (analyzed patients. For patient of group plitidepsin + dexamethasone the median overall survival could not be calculated due to follow-up short duration. The survival rates at 6 and 12 months are provided instead.
Measure: Number; unit: percentage patients
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Number analyzed (Participants) | 21 | 8
percentage patients
  OS at 6 months | 70 [5.1 to 31.8] | 76 [0 to 0]
  OS at 12 months | 53 | 61

ADVERSE EVENTS:
Description: 32 patients were treated with plitidepsin as single agent;afterwards 19 of them were treated with plitidepsin+dexamethasone combination.Therefore 32+19=51 is the no. patients at risk for plitidepsin and 19 is no. of patients at risk for dexamethasone
Arm/Group | Plitidepsin | Plitidepsin + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 32/51 | 11/19
Other Adverse Events (participants affected / at risk) | 51/51 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plitidepsin (N=51) | Plitidepsin + Dexamethasone (N=19)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy NOS (Cardiac disorders) | 1 | 0
Pulmonary oedema NOS (Cardiac disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection site cellulitis (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 0
Pyrexia (General disorders) | 7 | 3
Sudden death (General disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity NOS (Immune system disorders) | 0 | 1
Bronchitis acute NOS (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 7 | 2
Respiratory tract infection NOS (Infections and infestations) | 7 | 2
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Metabolic encephalopathy NOS (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute pre-renal failure (Renal and urinary disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 3 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Poor peripheral circulation (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plitidepsin (N=51) | Plitidepsin + Dexamethasone (N=19)
Anaemia NOS (Blood and lymphatic system disorders) | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiomegaly NOS (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhoea NOS (Gastrointestinal disorders) | 15 | 5
Dyspepsia (Gastrointestinal disorders) | 6 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hiccups (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 23 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 13 | 2
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 38 | 16
Injection site reaction NOS (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 7 | 4
Pain NOS (General disorders) | 2 | 2
Pyrexia (General disorders) | 20 | 3
Rigors (General disorders) | 3 | 1
Weakness (General disorders) | 3 | 2
Hepatic disorder NOS (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity NOS (Hepatobiliary disorders) | 4 | 0
Bronchitis NOS (Infections and infestations) | 1 | 1
Bronchitis acute NOS (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 1
Infection NOS (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Oral candidiasis (Infections and infestations) | 2 | 1
Respiratory tract infection NOS (Infections and infestations) | 7 | 3
Upper respiratory tract infection NOS (Infections and infestations) | 4 | 3
Urinary tract infection NOS (Infections and infestations) | 3 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Blood amylase increased (Investigations) | 3 | 1
Blood creatine phosphokinase (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Blood myoglobin increased (Investigations) | 0 | 1
Glucose urine present (Investigations) | 0 | 1
Weight decreased (Investigations) | 7 | 3
X-ray NOS chest abnormal (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 17 | 6
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 30 | 7
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 16 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 2
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 3 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Headache NOS (Nervous system disorders) | 6 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 3 | 1
Peripheral neuropathy NOS (Nervous system disorders) | 10 | 3
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Albuminuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 2
Haemoglobinuria (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 3 | 3
Renal failure NOS (Renal and urinary disorders) | 1 | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary vascular disorder NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep venous thrombosis NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
32 patients were treated with plitidepsin as single agent;afterwards 19 of them were treated with plitidepsin+dexamethasone combination.Therefore 32+19=51 is the no. patients at risk for plitidepsin and 19 is no. of patients at risk for dexamethasone

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other